CLINICAL TRIAL: NCT00631345
Title: Translating Research Into the Prevention of Diabetes Mellitus (TRIP DM)
Brief Title: Healthy Living Partnership to Prevent Diabetes
Acronym: HELP PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00000613; R18DK069901 (NIH); 1R18DK069901-01A2 (NIH)
Record Dates: First submitted 2008-03-05; First posted 2008-03-07 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Prediabetes; Obesity
Keywords: prediabetes; overweight; obesity; metabolic syndrome; community health worker
MeSH Terms: conditions — Prediabetic State; Obesity; Overweight; Metabolic Syndrome | interventions — Clinical Trials, Phase III as Topic; SDM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle (Experimental): This Group-Based Lifestyle Intervention (Phases 1 and 2) will be led by lay health counselors (LHCs). The 6-month Phase 1 includes weekly meetings on nutrition and physical activity, psychosocial factors related to health behaviors, and question and answer periods. The 18-month Phase 2 will consist of monthly group meetings and individual telephone contacts. Intervention participants who choose to participate in the study continuation (Phase 3) will be further randomized to receive either extended group or self-directed maintenance. Those who are randomized to receive Extended Group Maintenance (Phase 3) will continue attending monthly meetings; those who receive Self-Directed Maintenance (Phase 3) will no longer attend groups.
  Interventions: Behavioral: Group-Based Lifestyle Intervention (Phases 1 and 2); Behavioral: Self-Directed Maintenance (Phase 3); Behavioral: Extended Group Maintenance (Phase 3)
- Comparison (Other): The comparison condition exceeds the usual care provided to similar community members and is an individual education program that builds on an increased awareness of existing community resources. In the initial trial, these subjects will receive two individual sessions with the RD and a monthly newsletter. In the study continuation, comparison participants will receive biannual nutrition counseling and a monthly newsletter.
  Interventions: Other: Individual Education Program (All Phases)

INTERVENTIONS:
Behavioral: Group-Based Lifestyle Intervention (Phases 1 and 2) — This intervention involves a dietary weight loss program and an increase in caloric expenditure through moderate physical activity. The primary treatment objectives for the weight loss component of the intervention will be to decrease caloric intake in a nutritionally sound manner so as to produce a weight loss of approximately 0.3 kg per week for the first 6-months of treatment (Phase 1) for a total weight loss of 5-7%. During Phase 2 (months 7-24) participants will be encouraged to continue weight loss as long as their BMI does not fall below 20 kg/m2, but the primary focus will be on weight maintenance. The primary objective for the physical activity component of the intervention will be to promote an increase in home-based energy expenditure to an eventual goal of 180 min/week.
  Other Names: Community Health Worker-Led Intervention
  Arms: Lifestyle
Other: Individual Education Program (All Phases) — Comparison participants will receive two individual sessions with a nutritionist during the first 3 months. In these sessions, the RD will cover basic aspects of healthy eating and activity to support weight loss, discuss existing community resources and increased physical activity and weight loss. These participants will also receive a monthly newsletter on topics related to healthy lifestyle and will receive the lifestyle intervention manual and video series at the conclusion of their participation. These participants will be approached about the continuation at 24 months. If they agree to participate, these participants will continue to receive a monthly newsletter and will also receive biannual RD contacts.
  Other Names: Control
  Arms: Comparison
Behavioral: Self-Directed Maintenance (Phase 3) — Individuals from the lifestyle intervention group in the original HELP PD project who are randomized to self-directed maintenance will receive biannual nutrition counseling from the study RDs. In these sessions, the RD will cover basic aspects of transition from the group maintenance to individual maintenance, answer questions about healthy eating and activity to support weight loss, and discuss existing community resources that may fit the participants' needs as they attempt to maintain their weight loss, physical activity and dietary goals.
  Other Names: SDM
  Arms: Lifestyle
Behavioral: Extended Group Maintenance (Phase 3) — The extended group maintenance condition will consist of monthly CHW-led group meetings, monthly individual telephone contacts with the CHW, biannual RD contacts, and other contacts as needed. During Phase 3, the objectives for Phase 2 of the initial program will be continued. That is, participants who were successful at weight loss (≥ 7% of initial body weight) are encouraged to either maintain their weight loss or to advance towards their own personal goals. Participants who were not successful are encouraged to problem solve the reasons for lack of success. The groups will focus on maintaining the healthy behaviors that produced weight loss and/or problem solving to overcome barriers to weight loss.
  Other Names: EGM
  Arms: Lifestyle

SUMMARY:
The Healthy Living Partnership to Prevent Diabetes (HELP PD) is a 300-participant randomized trial designed to test the effectiveness of a lay-health counselor led community-based diabetes prevention program in reducing blood glucose in people at risk for developing diabetes mellitus.

DETAILED DESCRIPTION:
Social forces have promoted adverse behavioral patterns with respect to physical activity and nutrition resulting in the current epidemics of obesity, the metabolic syndrome and type 2 diabetes mellitus (DM). Results from clinical trials such as the Diabetes Prevention Program (DPP) have demonstrated a significant potential for prevention of type 2 DM through lifestyle interventions to promote physical activity, a healthy eating pattern and weight loss. Yet these approaches are not being applied in practice. In fact, whether these approaches can be successfully implemented in the community is an unanswered question. The Healthy Living Partnership to Prevent Diabetes (HELP PD) was designed to address this knowledge gap in a community setting. It incorporates key translations of prior research to enhance logistical and fiscal feasibility and long term dissemination, including the use of a group-based, rather than an individual-based, intensive lifestyle behavioral intervention employing professionals and community health workers (CHWs), and delivery of the intervention in the community setting via expansion of an existing Diabetes Education Program (DEP). The trial has been continued for an additional 5 years, and the primary goal of the continuation is to test the long-term glucose lowering effects of the HELP PD intervention by randomizing the lifestyle group to continued group maintenance or a self-directed maintenance condition and to follow the UC group for additional comparison purposes. Demonstrating the longer term effectiveness of HELP PD will represent a key step in establishing the value of this approach to translation of DM prevention into the community. This crucial evidence will be used to support reimbursement policy for DM prevention, dissemination of the HELP PD CHW approach and generalization to other behaviorally influenced chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Able to read/understand English at or above a level sufficient to comprehend recruitment and intervention materials
* BMI greater than or equal to 25 kg/m2 but less than 40 kg/m2
* Fasting blood glucose 95-125 mg/dl (inclusive)
* Willingness to Accept Randomization

Exclusion Criteria:

* Currently involved in a supervised program for weight loss
* Clinical history of DM, or newly diagnosed DM at screening
* Clinical history of cardiovascular disease (CVD) occurring within the past 6 months, including myocardial infarction, angina, coronary revascularization, stroke, TIA, carotid revascularization, peripheral arterial disease, and congestive heart failure
* Uncontrolled high blood pressure: BP > 160/100
* Pregnancy, breast feeding, or planning pregnancy within 2 years
* Other chronic disease likely to limit lifespan to less than 2-3 years, including any cancer requiring treatment in past 5 years except non-melanoma skin cancer
* Chronic use of medicine known to significantly affect glucose metabolism, e.g., corticosteroids
* Conditions/criteria likely to interfere with participation and acceptance of randomized assignment, including the following: inability/unwillingness to give informed consent, another household member already randomized to HELP PD, major psychiatric or cognitive problems (schizophrenia, dementia, self-reported active illegal substance or alcohol abuse), and participation in another research study that would interfere with HELP PD

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2007-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Fasting Glucose | Change from Baseline at 6, 12, 18, 24, 36, 42, 48, 54, 60, 66, 72 and 78 months from randomization
  Change in fasting glucose will be analyzed independently at 12 months (incorporating baseline and 6 month data) and will be used to report the average effect of the intervention during the first year. The analysis at 24 months (incorporating data from baseline, 18 and 24 months) will evaluate the long-term effects of the intervention by examining the average intervention effect during the second year of the intervention period.

SECONDARY OUTCOMES:
Weight Loss | Change from Baseline at 6, 12, 18, 24, 36, 42, 48, 54, 60, 66, 72 and 78 months from randomization
  Weight loss will be analyzed independently at 12 months (incorporating baseline and 6 month data) and will be used to report the average effect of the intervention during the first year. The analysis at 24 months (incorporating data from baseline, 18 and 24 months) will evaluate the long-term effects of the intervention by examining the average intervention effect during the second year of the intervention period.
Waist Circumference | Change from Baseline at 6, 12, 24, 36, 48, 60, and 72 months from randomization
  Waist circumference will be analyzed independently at 12 months (incorporating baseline and 6 month data) and will be used to report the average effect of the intervention during the first year. The analysis at 24 months (incorporating data from baseline, 18 and 24 months) will evaluate the long-term effects of the intervention by examining the average intervention effect during the second year of the intervention period.
Dietary Intake | Change from Baseline at 6, 12, 24, 36, 48, 60, and 72 months from randomization
  Usual dietary intake will be assessed using a food frequency questionnaire (FFQ) in web-format. This software will be administered during assessments at the GCRC by trained dieticians on the GCRC staff. In addition, diet will be monitored daily by intervention participants through completion of their diet and physical activity logs.
Physical Activity | Change from Baseline at 6, 12, 24, 36, 48, 60, and 72 months from randomization
  We will use the International Physical Activity Questionnaire to evaluate between group differences in physical activity, an internationally reliable and valid instrument for assessing physical activity. The IPAQ short form is a 7-item index that asks respondents the number of days per week and the amount of time per day spent in vigorous- and moderate-intensity activities and walking, during the seven days prior to the interview.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Z Vitolins, DrPH MPH RDN, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katula JA, Vitolins MZ, Rosenberger EL, Blackwell C, Espeland MA, Lawlor MS, Rejeski WJ, Goff DC. Healthy Living Partnerships to Prevent Diabetes (HELP PD): design and methods. Contemp Clin Trials. 2010 Jan;31(1):71-81. doi: 10.1016/j.cct.2009.09.002. Epub 2009 Sep 13. PMID 19758580
- [Background] Blackwell CS, Foster KA, Isom S, Katula JA, Vitolins MZ, Rosenberger EL, Goff DC Jr. Healthy Living Partnerships to Prevent Diabetes: recruitment and baseline characteristics. Contemp Clin Trials. 2011 Jan;32(1):40-9. doi: 10.1016/j.cct.2010.10.006. Epub 2010 Oct 23. PMID 20974289
- [Background] Katula JA, Blackwell CS, Rosenberger EL, Goff DC Jr; Healthy Living Partnerships to Prevent Diabetes Research Team. Translating diabetes prevention programs: implications for dissemination and policy. N C Med J. 2011 Sep-Oct;72(5):405-8. PMID 22416527
- [Background] Rosenberger Hale E, Goff DC, Isom S, Blackwell C, Whitt-Glover MC, Katula JA. Relationship of weekly activity minutes to metabolic syndrome in prediabetes: the healthy living partnerships to prevent diabetes. J Phys Act Health. 2013 Jul;10(5):690-8. doi: 10.1123/jpah.10.5.690. Epub 2012 Oct 4. PMID 23036940
- [Result] Katula JA, Vitolins MZ, Rosenberger EL, Blackwell CS, Morgan TM, Lawlor MS, Goff DC Jr. One-year results of a community-based translation of the Diabetes Prevention Program: Healthy-Living Partnerships to Prevent Diabetes (HELP PD) Project. Diabetes Care. 2011 Jul;34(7):1451-7. doi: 10.2337/dc10-2115. Epub 2011 May 18. PMID 21593290
- [Result] Katula JA, Vitolins MZ, Morgan TM, Lawlor MS, Blackwell CS, Isom SP, Pedley CF, Goff DC Jr. The Healthy Living Partnerships to Prevent Diabetes study: 2-year outcomes of a randomized controlled trial. Am J Prev Med. 2013 Apr;44(4 Suppl 4):S324-32. doi: 10.1016/j.amepre.2012.12.015. PMID 23498294
- [Result] Lawlor MS, Blackwell CS, Isom SP, Katula JA, Vitolins MZ, Morgan TM, Goff DC Jr. Cost of a group translation of the Diabetes Prevention Program: Healthy Living Partnerships to Prevent Diabetes. Am J Prev Med. 2013 Apr;44(4 Suppl 4):S381-9. doi: 10.1016/j.amepre.2012.12.016. PMID 23498303
- [Result] Bishop J, Irby MB, Isom S, Blackwell CS, Vitolins MZ, Skelton JA. Diabetes prevention, weight loss, and social support: program participants' perceived influence on the health behaviors of their social support system. Fam Community Health. 2013 Apr-Jun;36(2):158-71. doi: 10.1097/FCH.0b013e318282b2d3. PMID 23455686
- [Result] Beavers KM, Case LD, Blackwell CS, Katula JA, Goff DC Jr, Vitolins MZ. Effects of weight regain following intentional weight loss on glucoregulatory function in overweight and obese adults with pre-diabetes. Obes Res Clin Pract. 2015 May-Jun;9(3):266-73. doi: 10.1016/j.orcp.2014.09.003. Epub 2014 Oct 5. PMID 25293586
- [Result] Miller GD, Isom S, Morgan TM, Vitolins MZ, Blackwell C, Brosnihan KB, Diz DI, Katula J, Goff D. Effects of a community-based weight loss intervention on adipose tissue circulating factors. Diabetes Metab Syndr. 2014 Oct-Dec;8(4):205-11. doi: 10.1016/j.dsx.2014.09.003. Epub 2014 Oct 5. PMID 25293442
- [Result] Pedley CF, Case LD, Blackwell CS, Katula JA, Vitolins MZ. The 24-month metabolic benefits of the healthy living partnerships to prevent diabetes: A community-based translational study. Diabetes Metab Syndr. 2018 May;12(3):215-220. doi: 10.1016/j.dsx.2017.09.011. Epub 2017 Sep 23. PMID 28964720
- [Result] Vitolins MZ, Isom SP, Blackwell CS, Kernodle D, Sydell JM, Pedley CF, Katula JA, Case LD, Goff DC Jr. The healthy living partnerships to prevent diabetes and the diabetes prevention program: a comparison of year 1 and 2 intervention results. Transl Behav Med. 2017 Jun;7(2):371-378. doi: 10.1007/s13142-016-0447-z. PMID 27796775
- [Result] Vitolins MZ, Blackwell CS, Katula JA, Isom SP, Case LD. Long-term Weight Loss Maintenance in the Continuation of a Randomized Diabetes Prevention Translational Study: The Healthy Living Partnerships to Prevent Diabetes (HELP PD) Continuation Trial. Diabetes Care. 2019 Sep;42(9):1653-1660. doi: 10.2337/dc19-0295. Epub 2019 Jul 11. PMID 31296648